CLINICAL TRIAL: NCT05738499
Title: The Effectiveness and Mechanism of Character Strengths-based Structured Treatment and Education Programme on Rehabilitation of Stroke Patients
Brief Title: The Effectiveness and Mechanism of Character Strengths-based STEP Programme on Rehabilitation of Stroke Patients
Acronym: STEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, YAN Tingting, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00001052-22116
Record Dates: First submitted 2022-12-16; First posted 2023-02-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Intervention; Rehabilitation; Depression
Keywords: Stroke; Chronic illness management; Intervention; Post-stroke depression
MeSH Terms: conditions — Stroke; Depression | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSSTEP Group (Experimental): On the basis of routine post-stroke care, the CSSTEP programme was added for a total of three weeks. Each week includes one session course and three after-session strengths-based practicing activities. The names of the three sessions are: 1. Individualised education on character strengths and guidance on daily life skills in stroke; 2. Practicing activities on"three good things" of character strengths and physical rehabilitation training for stroke; 3. "New ways to use signature strengths" and secondary stroke prevention.
  Interventions: Other: Character strengths-based structured treatment and education programme (CSSTEP)
- Control Group (Placebo Comparator): On the basis of routine post-stroke care, the regular structured treatment and education programme will be comducted for a total of three weeks. Each week includes one session course of structured treatment and education programme.
  Interventions: Other: Structured treatment and education programme (STEP)

INTERVENTIONS:
Other: Character strengths-based structured treatment and education programme (CSSTEP) — This CSSTEP intervention included both psychological and educational contents, and the intervention type was psycho-educational intervention. The implementation process lasted for three weeks. CSSTEP mainly includes two main components. The first part is character strengths-based intervention. The second part is educational intervention, which is structured treatment and education programme for stroke patients. The two components were combined and optimized on the basis of theoritical and empirical evidences, and then this kind of complex intervention suitable for Chinese clinical stroke patients was obtained.
  Other Names: Psycho-educational intervention
  Arms: CSSTEP Group
Other: Structured treatment and education programme (STEP) — The STEP programme is aimed at the treatment needs of stroke patients, considering the education level and cultural background of patients, screening important health education content, and planning and grading of patients' education. The intervention consisted of three educational sessions, focusing on patients' daily life, post-stroke rehabilitation and secondary prevention.
  Other Names: Educational intervention
  Arms: Control Group

SUMMARY:
There is an urgent need for educational and psychological adjustment to stimulate the post-stroke patients' motivation to actively carry out rehabilitation. Studies have shown that interventions based on character strengths are widely used in chronic disease patients abroad, and have achieved the effect of improving the physical and mental health. However, research on individualized character strengths in stroke patient intervention is limited, and more clinical evidence is needed. This study is based on personality theory and the application of character strengths-based STEP programme (CSSTEP) in stroke patients. The investigators hypothesized that the CSSTEP programme could help stroke patients to improve mental state, cognitive function, and better gait performance, suffer from less post-stroke depression, enhance their post-stroke self-confidence.

DETAILED DESCRIPTION:
Post-stroke patients are often accompanied by different degrees of cognitive and language impairments. About 45% of the patients have persistent limb dysfunction, which leads to strong psychological stress reactions in patients, and negative emotions such as anxiety and depression are common. There is an urgent need for educational and psychological adjustment to stimulate the patient's motivation to actively carry out rehabilitation, so as to reduce negative emotions, enhance the patient's intrinsic motivation for rehabilitation, and reduce the patient's disability. Studies have shown that interventions based on character strengths are widely used in chronic disease patients abroad, and have achieved the effect of improving the physical and mental health of patients. However, research on individualized character strengths in stroke patient intervention is limited, and more clinical evidence is needed. This study is based on personality theory and the application of character strengths-based STEP programme (CSSTEP) in stroke patients. The investigators hypothesized that the CSSTEP programme could help stroke patients to improve mental state, cognitive function, and better gait performance, suffer from less post-stroke depression, enhance their post-stroke self-confidence. In addition, the investigators will use the application of CSSTEP in stroke care to provide a theoretical basis for a new personality direction for clinical psychological intervention, and provide new ideas and ideas for improving the stroke rehabilitation system and establishing a new personalized post-stroke intervention.

ELIGIBILITY:
Inclusion Criteria:

* ① Clinical diagnosis of stroke, CT or MRI diagnosis of cerebral infarction;
* ② Within 30 days after clinical diagnosis of acute stroke;
* ③ Age ≥18 years;
* ④ Basic cognition, learning ability and willingness, all vital signs were stable, no other serious complications and no history of mental illness;
* ⑤ Informed consent and cooperation.

Exclusion Criteria:

* ① Moderate or severe cognitive impairment (defined as mini-mental state examination score ≤20);
* ② Unstable vital signs, accompanied by severe heart, liver, renal insufficiency, respiratory failure and malignant tumors, unable to intervene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Depression at 1 month. Hamilton Depression Scale (HAMD-24) Scale | Baseline, Post-intervention within one week, One month after intervention
  This outcome will be measured by a specific scale/questionnaire, which is Hamilton Depression Scale (HAMD-24) Scale. Scores range from 0-52, higher scores mean worse outcome.

SECONDARY OUTCOMES:
Change from Baseline Self-esteem at 1 month. Rosenberg Self-esteem Scale (RSES) Scale | Baseline, Post-intervention within one week, One month after intervention
  This outcome will be measured by a specific scale/questionnaire, which is Rosenberg Self-esteem Scale (RSES) Scale. Scores range from 10-40, higher scores mean better outcome.
Change from Baseline Neurological function at 1 month. National Institutes of Health Stroke Scale (NIHSS) Scale | Baseline, Post-intervention within one week, One month after intervention
  This outcome will be measured by a specific scale/questionnaire, which is National Institutes of Health Stroke Scale (NIHSS) Scale. Scores range from 0-42, higher scores mean worse outcome.
Change from Baseline Cognitive function at 1 month. Mini-mental State Examination (MMSE) Scale | Baseline, Post-intervention within one week, One month after intervention
  This outcome will be measured by a specific scale/questionnaire, which is Mini-mental State Examination (MMSE) Scale. Scores range from 0-30, higher scores mean better outcome.
Change from Baseline Gait speed at 1 month | Baseline, Post-intervention within one week, One month after intervention
  This outcome will be measured by participants walking 10 metres with the camera filming the recording, recording the time taken and finally dividing the length of 10 metres by the time to obtain the average speed of the walk. The gait speed was measured in metres per second, which is m/sec. The results and data includes video of participants and gait speed.

CONTACTS AND LOCATIONS:
Overall Officials: Tingting YAN, PhD, Principal Investigator — Peking University
Locations (1):
- The Secind Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lou M, Ding J, Hu B, Zhang Y, Li H, Tan Z, Wan Y, Xu AD; Chinese Stroke Association Stroke Council Guideline Writing Committee. Chinese Stroke Association guidelines for clinical management of cerebrovascular disorders: executive summary and 2019 update on organizational stroke management. Stroke Vasc Neurol. 2020 Sep;5(3):260-269. doi: 10.1136/svn-2020-000355. Epub 2020 Jul 8. PMID 32641444
- [Background] Kakuda W. [Future directions of stroke rehabilitation]. Rinsho Shinkeigaku. 2020 Mar 31;60(3):181-186. doi: 10.5692/clinicalneurol.cn-001399. Epub 2020 Feb 26. Japanese. PMID 32101849
- [Background] Qian Z, Lv D, Lv Y, Bi Z. Modeling and Quantification of Impact of Psychological Factors on Rehabilitation of Stroke Patients. IEEE J Biomed Health Inform. 2019 Mar;23(2):683-692. doi: 10.1109/JBHI.2018.2827100. Epub 2018 Apr 16. PMID 29993937
- [Background] Rossignol S, Jones GM. Audio-spinal influence in man studied by the H-reflex and its possible role on rhythmic movements synchronized to sound. Electroencephalogr Clin Neurophysiol. 1976 Jul;41(1):83-92. doi: 10.1016/0013-4694(76)90217-0. PMID 58771
- [Background] Stahl B, Kotz SA, Henseler I, Turner R, Geyer S. Rhythm in disguise: why singing may not hold the key to recovery from aphasia. Brain. 2011 Oct;134(Pt 10):3083-93. doi: 10.1093/brain/awr240. Epub 2011 Sep 21. PMID 21948939
- [Background] Van Vleet TM, Robertson LC. Cross-modal interactions in time and space: auditory influence on visual attention in hemispatial neglect. J Cogn Neurosci. 2006 Aug;18(8):1368-79. doi: 10.1162/jocn.2006.18.8.1368. PMID 16859421
- [Background] Patel K, Watkins CL, Sutton CJ, Holland EJ, Benedetto V, Auton MF, Barer D, Chatterjee K, Lightbody CE. Motivational interviewing for low mood and adjustment early after stroke: a feasibility randomised trial. Pilot Feasibility Stud. 2018 Sep 25;4:152. doi: 10.1186/s40814-018-0343-z. eCollection 2018. PMID 30263147
- [Background] Watkins CL, Wathan JV, Leathley MJ, Auton MF, Deans CF, Dickinson HA, Jack CI, Sutton CJ, van den Broek MD, Lightbody CE. The 12-month effects of early motivational interviewing after acute stroke: a randomized controlled trial. Stroke. 2011 Jul;42(7):1956-61. doi: 10.1161/STROKEAHA.110.602227. Epub 2011 Jun 23. PMID 21700946
- [Background] Jokela M, Pulkki-Raback L, Elovainio M, Kivimaki M. Personality traits as risk factors for stroke and coronary heart disease mortality: pooled analysis of three cohort studies. J Behav Med. 2014 Oct;37(5):881-9. doi: 10.1007/s10865-013-9548-z. Epub 2013 Nov 8. PMID 24203126
- [Background] Afanasiev S, Aharon-Peretz J, Granot M. Personality type as a predictor for depressive symptoms and reduction in quality of life among stroke survivals. Am J Geriatr Psychiatry. 2013 Sep;21(9):832-9. doi: 10.1016/j.jagp.2013.04.012. Epub 2013 Jul 17. PMID 23871119
- [Background] Yan T, Chan CWH, Chow KM, Zheng W, Sun M. A systematic review of the effects of character strengths-based intervention on the psychological well-being of patients suffering from chronic illnesses. J Adv Nurs. 2020 Jul;76(7):1567-1580. doi: 10.1111/jan.14356. Epub 2020 Apr 7. PMID 32187708